CLINICAL TRIAL: NCT06811779
Title: Comparison of Effectiveness of Sodium Hypochlorite and Chlorhexidine Gluconate for Disinfection of Gutta Percha Cones
Brief Title: Comparison of Effectiveness of Disinfectants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Hira Amjad, Dr. Hafiza Hira Amjad, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Disinfection
Record Dates: First submitted 2025-01-19; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Root Canal Infection
Keywords: chemical disinfection; chlorhexidine gluconate; gutta percha; sodium hypochlorite
MeSH Terms: interventions — Sodium Hypochlorite; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Naocl group (Active Comparator): In this group, the Gp cones would be submerged in 5% naocl solution for 5 minutes and then tested for biofilm removal and eradication of inoculated microorganisms.
  Interventions: Drug: Sodium Hypochlorite
- chlorhexidine group (Active Comparator): In this group, the Gp cones would be submerged in 0.2% chlorhexidine solution for 5 minutes and then tested for biofilm removal and eradication of inoculated microorganisms.
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: Sodium Hypochlorite — Sodium hypochlorite used in 5% concentration for disinfection
  Arms: Naocl group
Drug: Chlorhexidine — Chlorhexidine 0.2% concentration for disinfection
  Arms: chlorhexidine group

SUMMARY:
This is a comparative experimental study to compare the efficacy of chemical disinfection agents , sodium hypochlorite and chlorhexidine gluconate in decontaminating gutta percha cones

DETAILED DESCRIPTION:
The study design is a comparative study which was done to compare the efficacy of chemical disinfection agents on decontaminating the gutta percha cones .

In this study, 124 standardized size-80 gutta-percha (GP) cones (Dentsply, Germany) were used to assess the efficacy of chemical disinfectants.

The cones were first sterilized using ethylene oxide to ensure baseline sterility. Following sterilization, 124 cones were allocated into two experimental groups (n = 62 each) for contamination.

group A . gp were immersed in 20ml of Enterococcus faecalis solution group B . gp were immersed in 20 ml of human saliva in patients undergoing root canal therapy

samples were incubated at 37°C for 72 hours to ensure uniform and thorough contamination

after incubation period cones were dried and divide into subgroups based on disinfectant agent applied .

The cones were immersed in disinfectant agent for 1 min and 10 min . Cones were dried again and immersed in brain heard infusion broth samples were again incubated at 37°C for 72 hours The presence of bacterial growth was determined by assessing turbidity in the broth, indicating viable microorganisms.

ELIGIBILITY:
Inclusion Criteria:

* healthy individual age between 20-40 patient needed root canal therapy

Exclusion Criteria:

* patient not willing to participate in study participants with systemic disease patients with neuromuscular disorder

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2024-03-24 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
effectiveness of disinfectants by assessing turbidity in broth using mann whitney test | 24 weeks
  Following disinfection, all gutta-percha (GP) cones were dried again with sterile gauze and placed individually into sterile test tubes containing 20 mL of fresh brain heart infusion (BHI) broth. The test tubes were incubated at 37°C for 72 hours. The presence of bacterial growth was determined by assessing turbidity in the broth, indicating viable microorganisms. Quantitative analysis of turbidity data was performed using the Mann-Whitney test and Kruskal-Wallis test to evaluate the effectiveness of the disinfectants across the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Hira Amjad, BDS, Principal Investigator — Armed Forces Institute of Dentistry
Locations (1):
- Armed Forces Institute of Dentistry, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No